CLINICAL TRIAL: NCT05228509
Title: Portal Vein Flow Velocity as a Screening Tool for Oesophageal Varices in Cirrhotic Patients
Acronym: Portalflow
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peter atef (Other)
Responsible Party: Sponsor-Investigator, Peter atef, Peter rizk, Assiut University
Organization: Assiut University (Other)
Other Study IDs: Patef
Record Dates: First submitted 2022-01-13; First posted 2022-02-08 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Cirrhosis Portal

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Portal vein flow velocity as screening tool for prediction of oesophageal varices in cirrhotic patient without upper endoscopy

DETAILED DESCRIPTION:
Portal vein flow velocity as screening tool for prediction of oesophageal varices in cirrhotic patient without upper endoscopy with its high cost & complications Using portal vein flow velocity and the relation between it & presence of oesophageal varices in cirrhotic patient & its efficacy as a primary tool for these cases

ELIGIBILITY:
Inclusion Criteria:

* cirrhotic patients with oesophageal varices
* cirrhotic patients without oesophageal varices

Exclusion Criteria:

* Patients with hepato-cellular carcinomas [HCCs], portal vein thrombosis, hepatic encephalopathy.
* Patients with positive HCV antibody, but without liver cirrhosis diagnostic criteria

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Cirrhotic patients with or without E
Sampling Method: Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2021-05-04 (Actual); Primary Completion 2024-12-02 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Using upper GIT endoscopy to detect the presence or absence of oesophageal varices | 3 years
  Non-invasive screening tool for esophageal varices:
  Aspartate aminotransferase-to-platelet ratio index (APRI) ... Doppler ultrasound of portal system Elastography both of liver and spleen... -Research outcome measures:
  a. Primary (main): Using upper GIT endoscopy to detect the presence or absence of oesophageal varices, and to detect the best and most available non- invasive predictor for it.

CONTACTS AND LOCATIONS:
Overall Officials: Peter At Munir, Master, Principal Investigator — Assiut University
Locations (2):
- Egypt (2):
  - 43, Asyut, Manfalout
  - Egypt .assiut.manfalout, Asyut, Manfalout